CLINICAL TRIAL: NCT02592798
Title: A Phase II Randomized, Placebo-Controlled, Double-Blind, Parallel Arms, Pilot Study to Evaluate the Efficacy and Safety of Intravenous Abatacept in Treatment Resistant Nephrotic Syndrome (Focal Segmental Glomerulosclerosis/ Minimal Change Disease)
Brief Title: Pilot Study to Evaluate the Safety and Efficacy of Abatacept in Adults and Children 6 Years and Older With Excessive Loss of Protein in the Urine Due to Either Focal Segmental Glomerulosclerosis (FSGS) or Minimal Change Disease (MCD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IM101-566; 2015-005450-36 (EudraCT Number)
Record Dates: First submitted 2015-10-29; First posted 2015-10-30 (Estimated); Results first posted 2021-03-05 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-02

CONDITIONS: Nephrotic Syndrome; Focal Segmental Glomerulosclerosis; Minimal Change Disease
MeSH Terms: conditions — Nephrotic Syndrome; Glomerulosclerosis, Focal Segmental; Nephrosis, Lipoid | interventions — Abatacept; Saline Solution; Glucose; Water

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Abatacept (Experimental): * Double Blind Periods 1 and 2 (DB1 and DB2): Abatacept IV administered on Day 1, 15, 29 and then every 28 days until the end of the Double Blind Period.
  * Open Label Period (OLE): Abatacept IV administered every 28 days
  Interventions: Drug: Abatacept
- Placebo (Placebo Comparator): * Double Blind Periods 1 and 2 (DB1 and DB2): Normal Saline or Dextrose 5% in Water (D5W) administer on Day 1, 15, 29 and then every 28 days until the end of the Double Blind Period.
  * Open Label Period (OLE): Abatacept IV administered every 28 days
  Interventions: Other: Normal Saline; Other: D5W

INTERVENTIONS:
Drug: Abatacept — Abatacept IV administered on Day 1, 15, 29 and then every 28 days
  Arms: Abatacept
Other: Normal Saline — Normal Saline administer on Day 1, 15, 29 and then every 28 days
  Arms: Placebo
Other: D5W — Dextrose 5% in Water (D5W) administered on Day 1, 15, 29 and then every 28 days
  Other Names: 5% Dextrose in Water
  Arms: Placebo

SUMMARY:
The purpose of this study is evaluate if abatacept is effective and safe in decreasing the level of protein loss in the urine in patients with excessive loss of protein in the urine (nephrotic syndrome) due to either focal segmental glomerulosclerosis (FSGS) or minimal change disease (MCD). Candidates must have a prior kidney biopsy with either diagnosis. Another kidney biopsy will not be required as part of the study. Candidates must have failed or be intolerant of prior therapy for their kidney disease. The failed or intolerant therapy must include corticosteroids and at least one other drug. Candidates can be adults and children over the age of 6. Abatacept will be administered by venous infusion every 4 weeks.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Male and female subjects ages ≥ 6 years
* Subjects resistant to corticosteroids, calcineurin inhibitors (cyclosporine and tacrolimus), sirolimus, mycophenolate mofetil (MMF), mycophenolic acid (MPA), or cyclophosphamide or intolerant to at least 2 of these
* UPCR ≥ 3 at screening
* FSGS or MCD confirmed by renal biopsy
* eGFR ≥ 45 for children and adults
* Concomitant use of angiotensin-converting-enzyme inhibitor (ACEi) or angiotensin receptor blocker (ARB) at stable doses for at least 2 weeks or have intolerance documented in the source documents maintained at the site

Exclusion Criteria:

* Kidney diseases other than FSGS or MCD
* Collapsing FSGS
* Systemic lupus erythematosus
* Diabetes mellitus, both type 1 and type 2
* Clinically significant congestive heart failure
* Post renal transplantation, including relapsing post-transplant FSGS
* Body mass index (BMI): > 40 in subjects ≥ 18 years of age and ≥ 99% percentile for subjects < 18 years of age

Other protocol defined inclusion/exclusion criteria may apply

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-03-09 (Actual); Primary Completion 2020-01-28 (Actual); Study Completion 2020-01-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (27):
- United States (27):
  - The University Of Alabama At Birmingham, Birmingham, Alabama
  - University of Alabama-Birmingham-Parent Account, Birmingham, Alabama
  - Los Angeles Biomedical Research Institute, Torrance, California
  - University Of Colorado Denver, Aurora, Colorado
  - Children's National Health System, Washington D.C., District of Columbia
  - University Of Miami Miller School Of Medicine, Miami, Florida
  - Nemours Childrens Hospital, Orlando, Florida
  - Emory University, Atlanta, Georgia
  - Loyola University Medical Center, Maywood, Illinois
  - NIH Clinical Center - NIDDK, Bethesda, Maryland
  - Boston Childrens Hospital, Boston, Massachusetts
  - Brigham And Women'S Hosp Inc., Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Childrens Mercy Hospital, Kansas City, Missouri
  - New York University Langone Medical Center, New York, New York
  - Columbia University Medical Center (Cumc), New York, New York
  - Levine Children's Hospital, Charlotte, North Carolina
  - Duke University, Durham, North Carolina
  - Cincinnati Children'S Hospital Medical Center, Cincinnati, Ohio
  - The Metro Health System, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - University Of Pennsylvania, Philadelphia, Pennsylvania
  - Local Institution, Pittsburgh, Pennsylvania
  - Renal Disease Research Institute, Dallas, Texas
  - University Of Texas Southwestern Medical Center, Dallas, Texas

REFERENCES:
- [Derived] Liu ID, Willis NS, Craig JC, Hodson EM. Interventions for idiopathic steroid-resistant nephrotic syndrome in children. Cochrane Database Syst Rev. 2025 May 8;5(5):CD003594. doi: 10.1002/14651858.CD003594.pub7. PMID 40337980
- [Derived] Azukaitis K, Palmer SC, Strippoli GF, Hodson EM. Interventions for minimal change disease in adults with nephrotic syndrome. Cochrane Database Syst Rev. 2022 Mar 1;3(3):CD001537. doi: 10.1002/14651858.CD001537.pub5. PMID 35230699
- [Derived] Hodson EM, Sinha A, Cooper TE. Interventions for focal segmental glomerulosclerosis in adults. Cochrane Database Syst Rev. 2022 Feb 28;2(2):CD003233. doi: 10.1002/14651858.CD003233.pub3. PMID 35224732
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 36 participants were randomized and treated.
Period: Double-Blind Period 1 (DB1)
Arm/Group | Abatacept | Placebo
Started | 17 | 19
Completed | 14 | 13
Not Completed | 3 | 6
Not completed — Pregnancy | 1 | 0
Not completed — No longer meeting study criteria | 0 | 1
Not completed — Lack of Efficacy | 1 | 3
Not completed — Adverse Event | 1 | 2
Period: Transition From DB1 to DB2
Arm/Group | Abatacept | Placebo
Started | 14 | 13
Completed | 11 | 11
Not Completed | 3 | 2
Not completed — Skipped DB2 and moved into subsequent OLE | 3 | 2
Period: Double-Blind Period 2 (DB2)
Arm/Group | Abatacept | Placebo
Started | 11 | 11
Completed | 6 | 9
Not Completed | 5 | 2
Not completed — Other reasons | 1 | 0
Not completed — Participant request to discontinue | 1 | 0
Not completed — No longer meeting study criteria | 1 | 0
Not completed — Lack of Efficacy | 1 | 2
Not completed — Adverse Event | 1 | 0
Period: Transition From DB2 to OLE
Arm/Group | Abatacept | Placebo
Started | 6 | 9
Completed | 5 | 9
Not Completed | 1 | 0
Not completed — Other reasons | 1 | 0
Period: Open Label Period (OLE)
Arm/Group | Abatacept | Placebo
Started (The starting pool of OLE period consists of participants who completed the Double-Blind Period + participants who escaped from DB1 and/or DB2 to OLE period) | 10 | 13
Completed | 6 | 4
Not Completed | 4 | 9
Not completed — Other reasons | 0 | 2
Not completed — Participant request to discontinue | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Lack of Efficacy | 3 | 5
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: * Double Blind Periods 1 and 2 (DB1 and DB2): Normal Saline or Dextrose 5% in Water (D5W) administered on Day 1, 15, 29 and then every 28 days until the end of the Double Blind Period.
  * Open Label Period (OLE): Abatacept IV administered every 28 days
- Total: Total of all reporting groups
Arm/Group | Abatacept | Placebo | Total
Number analyzed (Participants) | 17 | 19 | 36
Age, Continuous [Mean (Standard Deviation); unit: Years] | 22.5 (13.21) | 28.7 (19.35) | 25.8 (16.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 12 | 20
  Male | 9 | 7 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 7
  Not Hispanic or Latino | 15 | 14 | 29
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 3 | 7
  White | 13 | 14 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants in Renal Response at Day 113
Description: Renal Response is defined as the presence of all the following criteria:
  PROTEINURIA: Reduction of baseline urine protein/creatinine ratio (UPCR) of >= 50% and to less than 3.
  RENAL FUNCTION: No worsening of baseline estimated glomerular filtration rate (eGFR) defined as within normal range if normal at baseline or ≥ 75% baseline value if below normal at baseline.
Time Frame: From first dose to 113 days following first dose of the indicated period (113 days for Double-Blind Period, 226 days for Open Label Period)
Population: All treated participants with available measurements
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 17 | 19
Percent of Participants
  Double-Blind Period Day 113: number analyzed (Participants) | 13 | 13
  Double-Blind Period Day 113 | 0.0 [0.0 to 24.7] | 7.7 [0.2 to 36.0]
  Open Label Period Day 113: number analyzed (Participants) | 8 | 9
  Open Label Period Day 113 | 12.5 [0.3 to 52.7] | 33.3 [7.5 to 70.1]
Statistical Analysis 1: Comparison: Abatacept vs Placebo; Test type: Superiority; Mean Difference (Final Values) = -7.7, 95% CI 2-sided [-46.8 to 33.3] — Abatacept - Placebo for Double-Blind Period Day 113
Statistical Analysis 2: Comparison: Abatacept vs Placebo; Test type: Superiority; Mean Difference (Final Values) = -20.8, 95% CI 2-sided [-63.3 to 24.3] — Abatacept - Placebo for Open Label Period Day 113

2. Secondary Outcome: Mean Change From Baseline in Urine Protein/Creatinine Ratio (UPCR) at Day 113
Time Frame: From baseline (measured at day 1 of study) to 113 days following first dose administered in the indicated treatment period (113 days for Double-Blind Period, 226 days for Open Label Period)
Population: All treated participants with available measurements
Measure: Mean (Standard Error); unit: mg/mg
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 17 | 19
mg/mg
  Double-Blind Period Day 113: number analyzed (Participants) | 13 | 13
  Double-Blind Period Day 113 | 0.12 (0.5738) | -0.25 (0.7914)
  Open Label Period Day 113: number analyzed (Participants) | 8 | 8
  Open Label Period Day 113 | 1.98 (1.1598) | 0.02 (1.3049)
Statistical Analysis 1: Comparison: Abatacept vs Placebo; Test type: Superiority; Mean Difference (Final Values) = 0.37, 95% CI 2-sided [-1.6495 to 2.3855] — Abatacept - Placebo for Double-Blind Period Day 113
Statistical Analysis 2: Comparison: Abatacept vs Placebo; Test type: Superiority; Mean Difference (Final Values) = 1.95, 95% CI 2-sided [-1.7933 to 5.6954] — Abatacept - Placebo for Open Label Period Day 113

3. Secondary Outcome: Mean Change From Baseline in Serum Albumine at Day 113
Time Frame: From baseline (measured at day 1 of the study) to 113 days following first dose administered in the indicated treatment period (113 days for Double-Blind Period, 226 days for Open Label Period)
Population: All treated participants with available measurements
Measure: Mean (Standard Error); unit: g/dL
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 17 | 19
g/dL
  Double-Blind Period Day 113: number analyzed (Participants) | 11 | 12
  Double-Blind Period Day 113 | 0.08 (0.1016) | -0.05 (0.0892)
  Open Label Period Day 113: number analyzed (Participants) | 9 | 9
  Open Label Period Day 113 | 0.21 (0.1829) | 0.09 (0.2360)
Statistical Analysis 1: Comparison: Abatacept vs Placebo; Test type: Superiority; Mean Difference (Final Values) = 0.13, 95% CI 2-sided [-0.1483 to 0.4119] — Abatacept - Placebo for Double-Blind Period Day 113
Statistical Analysis 2: Comparison: Abatacept vs Placebo; Test type: Superiority; Mean Difference (Final Values) = 0.12, 95% CI 2-sided [-0.5107 to 0.7551] — Abatacept - Placebo for Open Label Period Day 113

4. Secondary Outcome: Percentage of Participants Achieving Complete Remission at Day 113
Description: Complete Remission is defined as the presence of all the following criteria:
  PROTEINURIA: Urine protein/creatinine ratio (UPCR) ≤ 0.3. RENAL FUNCTION: No worsening of baseline estimated glomerular filtration rate (eGFR) defined as within normal range if normal at baseline or ≥ 75% baseline value if below normal at baseline.
Time Frame: as for outcome 1
Population: All treated participants with available measurements
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 17 | 19
Percent of Participants
  Double-Blind Period Day 113: number analyzed (Participants) | 13 | 13
  Double-Blind Period Day 113 | 0.0 [0.0 to 24.7] | 0.0 [0.0 to 24.7]
  Open Label Period Day 113: number analyzed (Participants) | 8 | 9
  Open Label Period Day 113 | 12.5 [0.3 to 52.7] | 11.1 [0.3 to 48.2]
Statistical Analysis 1: Comparison: Abatacept vs Placebo; Test type: Superiority; Mean Difference (Final Values) = 1.4, 95% CI 2-sided [-44.7 to 44.7] — Abatacept - Placebo for Open Label Period Day 113

5. Secondary Outcome: Mean Change From Baseline in Patient Reported Outcomes Measurement Information System (PROMIS) at Day 113 - Adult Participants
Description: PROMIS was used to capture patient reported outcomes relevant to participants with nephrotic syndrome. Mean change from baseline is reported for the following measurements:
  Fatigue: Short From (SF) Fatigue v1.0 Adult 8a, composed of 8 questions, each one scored from 1 (Not at all) to 5 (Very much). Output presented as Total score, ranging from 8 (most desirable outcome) to 40 (least desirable outcome).
  Pain Interference: SF Pain Interference v1.0 Adult 8a, (measuring how much pain is interfering with daily activities). Composed of 8 questions, each one scored from 1 (Not at all) to 5 (Very much). Output presented as Total score, ranging from 8 (most desirable outcome) to 40 (least desirable outcome).
  Physical Function: SF Physical Function v1.2 Adult 8b, composed of 8 questions, each one scored from 1 (Without any difficulty) to 5 (Unable to do). Output presented as Total score, ranging from 8 (most desirable outcome) to 40 (least desirable outcome).
Time Frame: From baseline (measured at day 1 of study) to 113 days following first dose administered in the Double-Blind Period
Population: All treated participants with available measurements
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 9 | 11
Score on a scale
  Fatigue: number analyzed (Participants) | 8 | 8
  Fatigue | -5.56 (2.2907) | -4.87 (2.6125)
  Pain Interference: number analyzed (Participants) | 8 | 8
  Pain Interference | -4.88 (2.6395) | -1.18 (3.9785)
  Physical Function: number analyzed (Participants) | 8 | 8
  Physical Function | 0.78 (1.7350) | 1.77 (1.9346)
Statistical Analysis 1: Comparison: Abatacept vs Placebo; Test type: Superiority; Mean Difference (Final Values) = -0.69, 95% CI 2-sided [-8.1395 to 6.7645] — Abatacept - Placebo for Fatigue
Statistical Analysis 2: Comparison: Abatacept vs Placebo; Test type: Superiority; Mean Difference (Final Values) = -3.70, 95% CI 2-sided [-13.9402 to 6.5402] — Abatacept - Placebo for Pain interference
Statistical Analysis 3: Comparison: Abatacept vs Placebo; Test type: Superiority; Mean Difference (Final Values) = -1.00, 95% CI 2-sided [-6.5736 to 4.5736] — Abatacept - Placebo for Physical function

6. Secondary Outcome: Mean Change From Baseline in Patient Reported Outcomes Measurement Information System (PROMIS) at Day 113 - Pediatric Participants
Description: PROMIS was used to capture patient reported outcomes relevant to participants with nephrotic syndrome. Mean change from baseline is reported for the following measurements:
  Fatigue: Short From (SF) Fatigue v1.0 Peds 10a, composed of 10 questions, each one scored from 0 (Never) to 4 (Almost Always). Output presented as Total score, ranging from 0 (most desirable outcome) to 40 (least desirable outcome).
  Pain Interference: SF Pain Interference v1.0 Peds 8a, ( measuring how much pain is interfering with daily activities). Composed of 8 questions, each one scored from 0 (Never) to 4 (Almost always). Output presented as Total score, ranging from 0 (most desirable outcome) to 32 (least desirable outcome).
  Mobility: SF Physical Function-Mobility v1.0 Peds 8a, composed of 8 questions, each one scored from 0 (Not able to do) to 4 (With no trouble). Output presented as Total score, ranging from 0 (least desirable outcome) to 32 (most desirable outcome).
Time Frame: From baseline (measured at day 1 of study) to 113 days following first dose administered in the Double-Blind Period
Population: All treated participants with available measurements
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 8 | 8
Score on a scale
  Fatigue: number analyzed (Participants) | 4 | 5
  Fatigue | 6.43 (6.7142) | -6.02 (3.6526)
  Pain Interference: number analyzed (Participants) | 4 | 5
  Pain Interference | 5.70 (3.9781) | -1.44 (1.9180)
  Mobility: number analyzed (Participants) | 4 | 5
  Mobility | 0.80 (3.5007) | 1.68 (3.1905)
Statistical Analysis 1: Comparison: Abatacept vs Placebo; Test type: Superiority; Mean Difference (Final Values) = 12.45, 95% CI 2-sided [-4.5950 to 29.4850] — Abatacept - Placebo for Fatigue
Statistical Analysis 2: Comparison: Abatacept vs Placebo; Test type: Superiority; Mean Difference (Final Values) = 7.14, 95% CI 2-sided [-2.5917 to 16.8717] — Abatacept - Placebo for Pain interference
Statistical Analysis 3: Comparison: Abatacept vs Placebo; Test type: Superiority; Mean Difference (Final Values) = -0.88, 95% CI 2-sided [-12.1068 to 10.3468] — Abatacept - Placebo for Mobility

7. Secondary Outcome: Number of Participants Experiencing Adverse Events
Description: This outcome describes the number of participants experiencing various types of any grade Adverse Events (AEs).
  The Cumulative Abatacept Safety Period starts at the time of the first dose of Abatacept (either in the Double-Blind Period or in the Open Label Period) and lasts 56 days after the last dose of Abatacept
Time Frame: From first dose in the indicated period to 56 days following last dose in the indicated period (169 days for the Double-Blind Period, up to 337 days for the Cumulative Abatacept Safety Period)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Groups:
- Abatacept During Double-Blind Period: Abatacept IV administered on Day 1, 15, 29 and then every 28 days until the end of the Double Blind Period.
- Placebo During Double-Blind Period: Normal Saline or Dextrose 5% in Water (D5W) administer on Day 1, 15, 29 and then every 28 days until the end of the Double Blind Period.
- Abatacept During Cumulative Abatacept Safety Period: Any participants receiving at least 1 dose of Abatacept, starting either in the Double-Blind Period or in the Open Label Period
Arm/Group | Abatacept During Double-Blind Period | Placebo During Double-Blind Period | Abatacept During Cumulative Abatacept Safety Period
Number analyzed (Participants) | 17 | 19 | 32
Participants
  Adverse Events (AEs) | 13 | 15 | 26
  Serious Adverse Events (SAEs) | 5 | 4 | 10
  AEs leading to discontinuation | 1 | 2 | 2
  Deaths | 0 | 0 | 0

8. Secondary Outcome: Number of Participants Experiencing Adverse Events of Special Interest
Description: Number of participants experiencing various types of Adverse Events of interest, including infections, malignancies, autoimmune disorders, and infusional related reactions.
Time Frame: From first dose on day 1 to 56 days following last dose (approximately 330 days)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 17 | 19
Participants
  Peri-infusional Adverse Event (AE) | 6 | 3
  AE within 24 hours of Infusion | 8 | 9
  Malignancies | 0 | 0
  Infections/Infestations | 12 | 10
  Autoimmune disorders | 0 | 1

9. Secondary Outcome: Percentage of Participants With Positive Antibody Response Relative to Baseline
Description: A positive response relative to baseline is defined as a positive response at a post-baseline visit that has a titer value greater than the positive baseline titer value. If the baseline titer is missing or negative, any post-baseline positive titer value is considered a positive response relative to baseline.
  Immunogenicity response is presented as the total of immunogenicity response for "CTLA4 and possibly Ig" and "Ig and/or Junction Region".
Time Frame: From baseline (day 1) to 168 days following last dose (up to 15 months). Results at day 113 from first dose, day 56, day 84 and day 168 after last dose are presented
Population: All treated participants with available measurements
Measure: Number; unit: Percent of Participants
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 17 | 19
Percent of Participants
  Day 113 from first dose: number analyzed (Participants) | 14 | 12
  Day 113 from first dose | 7.1 | 0.0
  Day 56 from last dose: number analyzed (Participants) | 5 | 3
  Day 56 from last dose | 40.0 | 66.7
  Day 84 from last dose: number analyzed (Participants) | 7 | 3
  Day 84 from last dose | 28.6 | 66.7
  Day 168 from last dose: number analyzed (Participants) | 6 | 4
  Day 168 from last dose | 16.7 | 25.0

10. Secondary Outcome: Minimum Blood Plasma Concentration (Cmin) of Abatacept - Adult Participants
Time Frame: From first dose to 113 days after first dose in the Double Blind Period. Data collected on day 15, day 29, day 57, day 85 and day 113
Population: All adult participants receiving Abatacept during the Double Blind Period with available measurements
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 17 | 19
ug/mL
  Day 15: number analyzed (Participants) | 9 | 0
  Day 15 | 7.613 (63.7) |
  Day 29: number analyzed (Participants) | 8 | 0
  Day 29 | 12.274 (86.7) |
  Day 57: number analyzed (Participants) | 9 | 0
  Day 57 | 3.641 (66.5) |
  Day 85: number analyzed (Participants) | 7 | 0
  Day 85 | 4.101 (52.7) |
  Day 113: number analyzed (Participants) | 7 | 0
  Day 113 | 2.786 (68.2) |

11. Secondary Outcome: Minimum Blood Plasma Concentration (Cmin) of Abatacept - Pediatric Participants
Time Frame: as for outcome 10
Population: All pediatric participants receiving Abatacept during the Double Blind Period with available measurements
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 17 | 19
ug/mL
  Day 15: number analyzed (Participants) | 8 | 0
  Day 15 | 2.829 (116.4) |
  Day 29: number analyzed (Participants) | 7 | 0
  Day 29 | 2.588 (138.7) |
  Day 57: number analyzed (Participants) | 8 | 0
  Day 57 | 0.504 (143.2) |
  Day 85: number analyzed (Participants) | 5 | 0
  Day 85 | 1.617 (123.5) |
  Day 113: number analyzed (Participants) | 6 | 0
  Day 113 | 0.990 (163.1) |

12. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of Abatacept
Time Frame: Day 85 after first dose in the Double Blind Period
Population: All participants receiving Abatacept during the Double Blind Period with available measurements
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 17 | 19
ug/mL
  Adult participants: number analyzed (Participants) | 7 | 0
  Adult participants | 200.46 (43.9) |
  Pediatric participants: number analyzed (Participants) | 6 | 0
  Pediatric participants | 174.65 (30.0) |

13. Secondary Outcome: Area Under the Serum Concentration Time Curve Over a Dosing Interval (AUC(TAU)) of Abatacept
Time Frame: From Day 85 to Day 113 in the Double Blind Period
Population: All participants receiving Abatacept during the Double Blind Period with available measurements
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug*h/mL
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 17 | 19
ug*h/mL
  Adult participants: number analyzed (Participants) | 7 | 0
  Adult participants | 20394.83 (44.3) |
  Pediatric participants: number analyzed (Participants) | 4 | 0
  Pediatric participants | 18282.50 (41.9) |

14. Secondary Outcome: Time to Reach Peak Serum Concentration (Tmax(h)) of Abatacept
Time Frame: Day 85 after first dose in the Double Blind Period
Population: All participants receiving Abatacept during the Double Blind Period with available measurements
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 17 | 19
Hours
  Adult participants: number analyzed (Participants) | 7 | 0
  Adult participants | 0.883 (0.242) |
  Pediatric participants: number analyzed (Participants) | 6 | 0
  Pediatric participants | 0.589 (0.285) |

ADVERSE EVENTS:
Time Frame: From first dose to 100 days following administration of last dose (approximately 1 year)
Groups:
- Abatacept During Double-Blind Period 1 (DB1); Abatacept During Double-Blind Period 2 (DB2): Abatacept IV administered on Day 1, 15, 29 and then every 28 days until the end of the Double Blind Period.
- Placebo During Double-Blind Period 1 (DB1); Placebo During Double-Blind Period 2 (DB2): Normal Saline or Dextrose 5% in Water (D5W) administered on Day 1, 15, 29 and then every 28 days until the end of the Double Blind Period.
- Abatacept During Open Label Period (OLE): Abatacept IV administered every 28 days
Arm/Group | Abatacept During Double-Blind Period 1 (DB1) | Placebo During Double-Blind Period 1 (DB1) | Abatacept During Double-Blind Period 2 (DB2) | Placebo During Double-Blind Period 2 (DB2) | Abatacept During Open Label Period (OLE)
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/19 | 0/11 | 0/11 | 0/23
Serious Adverse Events (participants affected / at risk) | 5/17 | 4/19 | 0/11 | 2/11 | 6/23
Other Adverse Events (participants affected / at risk) | 13/17 | 15/19 | 7/11 | 8/11 | 16/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abatacept During Double-Blind Period 1 (DB1) (N=17) | Placebo During Double-Blind Period 1 (DB1) (N=19) | Abatacept During Double-Blind Period 2 (DB2) (N=11) | Placebo During Double-Blind Period 2 (DB2) (N=11) | Abatacept During Open Label Period (OLE) (N=23)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 0
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Periorbital swelling (Eye disorders) | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Lip swelling (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0 | 0
Generalised oedema (General disorders) | 2 | 0 | 0 | 0 | 1
Oedema (General disorders) | 2 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 2
Fluid overload (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 2 | 0 | 1 | 1
Nephrotic syndrome (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0
Renal disorder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Renal tubular necrosis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Abatacept During Double-Blind Period 1 (DB1) (N=17) | Placebo During Double-Blind Period 1 (DB1) (N=19) | Abatacept During Double-Blind Period 2 (DB2) (N=11) | Placebo During Double-Blind Period 2 (DB2) (N=11) | Abatacept During Open Label Period (OLE) (N=23)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Nephrogenic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Splenomegaly (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 1 | 0 | 0 | 0
Middle ear effusion (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 2 | 0 | 0 | 0 | 0
Eye inflammation (Eye disorders) | 0 | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 4 | 3 | 0 | 1 | 3
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 2 | 1 | 1 | 4
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 5 | 2 | 0 | 0 | 3
Chest pain (General disorders) | 1 | 0 | 0 | 0 | 0
Complication associated with device (General disorders) | 0 | 0 | 1 | 0 | 0
Energy increased (General disorders) | 1 | 0 | 0 | 0 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 2
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 1
Feeling cold (General disorders) | 0 | 1 | 0 | 0 | 0
Malaise (General disorders) | 0 | 1 | 0 | 0 | 0
Nodule (General disorders) | 0 | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0 | 1
Oedema (General disorders) | 4 | 2 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 3 | 0 | 0 | 1
Pain (General disorders) | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 2 | 0 | 0 | 4
Swelling (General disorders) | 0 | 0 | 0 | 1 | 1
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Ear infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Furuncle (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Gastrointestinal viral infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Pulpitis dental (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1 | 1 | 4
Viral pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Heat cramps (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Blood albumin decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 2 | 0 | 1 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 1 | 0
Blood triglycerides increased (Investigations) | 0 | 0 | 1 | 1 | 0
Influenza A virus test positive (Investigations) | 0 | 0 | 1 | 0 | 0
Respiratory syncytial virus test positive (Investigations) | 0 | 1 | 0 | 0 | 0
Weight increased (Investigations) | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0
Dizziness (Nervous system disorders) | 3 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 5 | 1 | 2 | 2
Visual field defect (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 3
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 1 | 1
Panic attack (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Nephrotic syndrome (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Amenorrhoea (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Polymenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 2
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Alopecia areata (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 1
Skin lesion inflammation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 2 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Amendment 02 of the Clinical Protocol (18 April 2018) modified the study design, so that the Double-Blind Period (DB) would not include anymore 2 consecutive periods (DB1 and DB2). However, for transparency and completeness reasons, in the Participant Flow and Adverse Events sections data about DB1 and DB2 are reported separately.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2018-04-18): https://cdn.clinicaltrials.gov/large-docs/98/NCT02592798/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-06): https://cdn.clinicaltrials.gov/large-docs/98/NCT02592798/SAP_001.pdf